CLINICAL TRIAL: NCT04859647
Title: Client-led Online Therapy for People Diagnosed With Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Kadie-Charelle Roberts, Trainee Clinical Psychologist, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 288776
Record Dates: First submitted 2021-04-07; First posted 2021-04-26 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Bipolar Spectrum Disorder
Keywords: Novel intervention; Psychological therapy; Online therapy; Client-led; Method of levels; Case Series
MeSH Terms: interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapy Intervention (Other): Method of Levels Therapy Intervention - Clients will choose how many sessions to attend during the 6 months therapy window. Clients will also choose how often to attend sessions and the duration of each session.
  Interventions: Other: Method of Levels Therapy

INTERVENTIONS:
Other: Method of Levels Therapy — MOL is a flexible, client-led psychological therapy that allows people to talk freely about important problems and life goals.
  Other Names: Psychological Therapy; Talking Therapy; Psychotherapy

SUMMARY:
The study aims to investigate the use of Method of Levels therapy (MOL) delivered online via videoconferencing for people who have received a diagnosis of a bipolar spectrum disorder. People are typically offered medication and talking therapies aimed at reducing symptoms and managing relapse. Research shows, however, that people tend to report reasons for distress other than symptoms and prioritise a fulfilling, purposeful life over remaining relapse- free. Having choice and control over treatment have been identified as important aspects of recovery in bipolar disorder.

MOL is a flexible, client-led psychological therapy that allows people to talk freely about important problems and life goals. MOL has already been applied to a range of mental health difficulties with promising results.

The aims of the study are to:

* Investigate whether it is feasible to deliver MOL online to people with a bipolar spectrum disorder
* Investigate whether MOL delivered online is an acceptable psychological intervention for people with a bipolar spectrum disorder
* Identify the elements of therapy that people want choice over and the impact and importance of these elements
* Determine whether there is a link between how much control over therapy people perceive themselves to have and the degree to which they generate new perspectives, thoughts and insights into their problems.

The current study will aim to recruit a minimum of 12 participants with a diagnosis of Bipolar Spectrum Disorder to account for 30% attrition (a conservative estimate based on reported attrition rates for published studies evaluating Cognitive Behavioural Therapy (CBT) for Bipolar Disorder). Therefore, the study aims to retain 8 participants for completion of the study. This is considered feasible in the available timeframe as recruitment will adopt a broad strategy. Participants will be offered MOL sessions online for up to six months. Potential participants will choose how many sessions to have, when to attend and what to talk about. Investigators will consider how many participants chose to take part and remain in the study to the end. The investigators will also ask participants about their experiences of the intervention and any changes participants may have noticed via feedback questionnaires and an interview.

DETAILED DESCRIPTION:
Bipolar spectrum disorder (previously known as manic depression) is a diagnostic term used to describe experiences of extreme, and sometimes enduring, fluctuations in mood that interfere with a person's life or cause significant distress. Individuals diagnosed with bipolar disorder experience periods of depressed mood and periods of elevated or irritable mood. In many cases, this amounts to clinical depression, or mania that entails hospital admission. Periods of mood fluctuation usually involve extreme changes to usual thinking and behaviour. During a period of depression people might feel hopeless and suicidal, withdraw from social activities and have difficulty functioning, resulting in a neglect of self-care and basic needs. During mania people might experience delusional beliefs, become highly distractible and prone to engaging in high-risk activities such as excessive spending or drug-taking. Both mood states can result in significant impairment in work, social or daily functioning and may result in hospitalisation.

Many people with a diagnosis of a bipolar spectrum disorder experience multiple relapses, causing them significant long-term disability. Meeting the needs of this client group can pose a real challenge for services given the complexity of fluctuating mood states, high levels of impulsivity and associated risk, and additional difficulties that people can also experience (such as anxiety and trauma).

Current guidelines recommend that people who have received a diagnosis of a bipolar spectrum disorder are offered an evidence-based psychological intervention as well as medication. These interventions are typically time-limited and guided by a specific manual with emphasis on alleviating symptoms and relapse prevention. The quality of the evidence supporting such interventions has been questioned. There has also been doubt cast on the effectiveness of these interventions.

Treatment adherence is also considered suboptimal, with relatively high drop-out rates. Access to talking therapies for those with complex needs has been described as 'notoriously poor'. People diagnosed with a bipolar spectrum disorder often report reasons for distress other than symptoms and prioritise a fulfilling, purposeful life over remaining relapse-free. Talking freely to a caring, approachable therapist is valued, as are interventions that facilitate control over aspects of life beyond mood. Recovery is achievable when people are empowered to follow a self- determined path, take ownership and confront longstanding problems.

Recent advances in cognitive therapy have departed from traditional relapse prevention to offer a theory-based approach that helps people understand their individual experience of bipolar spectrum disorder and target current problems and control over life goals (rather than focusing on controlling swings). Although patients perceived the intervention to be beneficial, a trial did not find significant improvement compared to treatment as usual. Patients wanted more sessions and greater flexibility in scheduling, and many reported problems beyond their diagnosis.

More client-led approaches that are not tied to the specific diagnosis could better suit the therapeutic needs of people diagnosed with a bipolar spectrum disorder. One such approach is Method of Levels (MOL); an application of Perceptual Control Theory (PCT). PCT proposes that distress arises when people strive to achieve conflicting goals. People are typically able to resolve the conflict and re-establish control through a natural trial-and- error process. This process becomes disrupted when people remain unaware of the conflict. The questioning approach of MOL therefore aims to help people develop greater awareness of important goals and conflicts, and consider problems from new perspectives, thus generating their own solutions. For example, a client diagnosed with a bipolar spectrum disorder may work through their dilemma over whether to devote their life to their success as a creative writer, or to their relationship with their family; or they may be struggling between disclosing a past traumatic assault to the police to get justice, or to keep the experience to themselves for fear of reprisal or ridicule.

MOL has potential advantages over existing psychological approaches; it offers flexible, client-led appointment scheduling, it can be applied to a range of problems causing distress, treatment is tailored to individual needs, and it aims to provide people with more choice and control over the interventions they receive.

Perceived control, identified as a key mechanism of psychological change in MOL therapy, has been shown to contribute to decreased levels of overall distress. Perceived control has been linked to an increased awareness of the problem, an ability to talk freely and develop problem resolution. Client perceptions of control are closely related to their perceptions of helpfulness; both factors have been associated with effectiveness of therapy.

MOL has shown promising results in a variety of settings, including primary care, secondary care and inpatient hospital settings. It has been applied to a range of problems, including complex mental health problems such as psychosis.

Remote delivery of MOL via videoconferencing could further improve the level of flexibility and control offered to patients. There is promising evidence that video therapy can be clinically effective and acceptable to patients; when managed well it can also reduce costs for health services. Delivery via videoconferencing fits in with the flexible, client-led ethos of MOL, and is highly relevant given the current COVID-19 pandemic and associated restrictions on face to face therapy. MOL is interaction based, with no reliance on written information; it could be offered remotely from a practical perspective. It would seem that MOL has the potential to meet the needs of those who have received a diagnosis of a bipolar spectrum disorder, particularly when offered via videoconferencing.

To date, there have been no published studies evaluating MOL as a potential intervention for bipolar spectrum disorder. The feasibility and acceptability of offering MOL via videoconferencing has not yet been established. The proposed study therefore aims to evaluate the feasibility and acceptability of MOL, delivered via videoconferencing, as an intervention for people with a diagnosis of a bipolar spectrum disorder.

Given the importance of perceived control within therapy, the study also aims to provide an opportunity to explore the elements of therapy that people want choice over and the impact and importance of these elements. Considering the effectiveness of the intervention (in terms of reduction of distress and improvements in functioning and goal attainment) is a secondary aim of the study. An additional secondary aim is to determine whether there is a link between how much control over therapy participants perceive themselves to have and the degree to which they generate new perspectives, thoughts and insights.

The results of the study could help to inform future research into the clinical effectiveness of MOL for those with a diagnosis of a bipolar spectrum disorder, as well as the most effective methods of delivery for this therapy. It could also help inform developments in psychological therapies more broadly by considering the importance people place on perceiving themselves to have more choice and to feel in control during therapy and the impact this has on psychological change and overall wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18 years and over
* Individuals with a diagnosis of Bipolar Spectrum Disorder.
* People accessing services or third sector agencies and/ or living in England.
* Access to personal use of technology is required for online therapy.

Exclusion Criteria:

* People presenting with extreme risk to self or others and engaging in active suicidal thoughts and/or behaviours.
* Problems of an organic nature, such as a brain injury or learning disability that might affect cognitive functioning.
* People already receiving a talking therapy for their difficulties
* People unable to speak/ understand sufficient English.
* Anyone already receiving talking therapy at the time of enrolment
* Anyone with a diagnosis of schizophrenia, schizoaffective disorder, primary substance misuse (mood swings caused purely by substance misuse), or psychosis outside of mood episodes or current episode of mania.
* People who do not have access to the internet and a video calling device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of Study through recruitment of participants | Through study completion, up to 6 months
  Feasibility will be measured by the proportion of eligible people recruited (based on the number of eligible referrals who chose to participate). These multiple measurements of feasibility will be combined to calculate an overall percentage of completion. Based on a recent trial with this client group, the percentage of eligible people needed to be recruited, remain in the study and complete the outcome measures to signal feasibility will be set conservatively at 50 percent. The number of sessions cancelled or terminated prematurely due to technical problems will also be considered.
Feasibility of Study through retention of participants | Through study completion, up to 6 months
  Feasibility will be measured by participant retention rates (the number of people that remain in the study until the end of the study). These multiple measurements of feasibility will be combined to calculate an overall percentage of completion. Based on a recent trial with this client group, the percentage of eligible people needed to be recruited, remain in the study and complete the outcome measures to signal feasibility will be set conservatively at 50 percent. The number of sessions cancelled or terminated prematurely due to technical problems will also be considered.
Feasibility of Study through data completion | Through study completion, up to 6 months
  Feasibility will be measured by the proportion of data completion (the number of outcome measures completed by participants during the study). These multiple measurements of feasibility will be combined to calculate an overall percentage of completion. Based on a recent trial with this client group, the percentage of eligible people needed to be recruited, remain in the study and complete the outcome measures to signal feasibility will be set conservatively at 50 percent. The number of sessions cancelled or terminated prematurely due to technical problems will also be considered.
Acceptability of Intervention through written feedback | Through study completion, up to 6 months
  The key measure of acceptability will be a content analysis of written feedback comments. Feedback relating to quality of connection, audio, and video, and any impact of technological problems will also be considered. Descriptive statistics for the number of sessions attended, cancelled, not attended without prior notice, and the length of sessions will be provided. Where participants cancel or fail to attend a prearranged session, drop out of the study, or book few or no sessions, attempts will be made to ascertain the reasons. The collective data will determine whether the intervention would be considered acceptable by participants. A post-treatment retention rate of at least 75 percent would be considered to indicate acceptability in this study.

SECONDARY OUTCOMES:
Working Alliance Inventory - Short Version Revised (WAI-SR; Paap & Dijkstra, 2017). | During the Intervention, up to 26 weeks
  Mean scores from the WAI-SR will also be presented as measures of acceptability. The 12-item self report scale aims to measure key aspects of therapeutic alliance; agreement regarding the goals of treatment, the tasks to achieve goals and the quality of the client-therapist bond. The higher the scores on the WAI-SR, the greater the degree of acceptability.

OTHER OUTCOMES:
The Active Involvement Scale (AIS) - A measure of client experience and key perceptions of therapy | During the intervention, up to 6 months
  The Active Involvement Scale (AIS) - a 5 item feedback questionnaire devised specifically to capture and focus on the participant's experience of the therapy session; their ability to talk openly about their problem and their perception of what they believe to be the key elements of the therapy, and how these are experienced. Each item scale ranges from 0-10, with 10 being the highest score, and therefore indicates a high level of perceived control and choice. It is anticipated that 50 percent of scores above 5 on the AIS would indicate perceived control during therapy and reflect changes in perceived distress during the course of treatment. Total scores range from 0-40.
Perceived choice and control in therapy | During the intervention, up to 3 months
  Qualitative interviews will be the most significant indicator of perceived choice and control during therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Kadie Roberts, Principal Investigator — Trainee Clinical Psychologist, The University of Manchester
Locations (1):
- The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The findings of this study will be written up as a Doctorate level thesis, which will be available at the University of Manchester library. Articles will also be submitted for publication in peer reviewed scientific journals. The research team will offer to feedback the results of the study to the National Health Service (NHS) clinical teams and Charities that were involved in the recruitment of participants. This will be done via a written lay summary. Participants can also request a written summary or copy of any published articles.
  No identifiable personal data will be published when writing up the findings of this study. Individual participants will not be identifiable through the combination of data being published.

REFERENCES:
- [Background] Searson R, Mansell W, Lowens I, Tai S. Think Effectively About Mood Swings (TEAMS): a case series of cognitive-behavioural therapy for bipolar disorders. J Behav Ther Exp Psychiatry. 2012 Jun;43(2):770-9. doi: 10.1016/j.jbtep.2011.10.001. Epub 2011 Oct 15. PMID 22104659
- [Background] Mansell W, Tai S, Clark A, Akgonul S, Dunn G, Davies L, Law H, Morriss R, Tinning N, Morrison AP. A novel cognitive behaviour therapy for bipolar disorders (Think Effectively About Mood Swings or TEAMS): study protocol for a randomized controlled trial. Trials. 2014 Oct 24;15:405. doi: 10.1186/1745-6215-15-405. PMID 25344393
- [Background] Gaffney H, Mansell W, Tai S. Conversational Agents in the Treatment of Mental Health Problems: Mixed-Method Systematic Review. JMIR Ment Health. 2019 Oct 18;6(10):e14166. doi: 10.2196/14166. PMID 31628789
- [Background] Griffiths R, Mansell W, Carey TA, Edge D, Emsley R, Tai SJ. Method of levels therapy for first-episode psychosis: rationale, design and baseline data for the feasibility randomised controlled Next Level study. BJPsych Open. 2018 Aug 14;4(5):339-345. doi: 10.1192/bjo.2018.44. eCollection 2018 Sep. PMID 30140445
- [Background] Davenport K, Hardy G, Tai S, Mansell W. Individual experiences of psychological-based interventions for bipolar disorder: A systematic review and thematic synthesis. Psychol Psychother. 2019 Dec;92(4):499-522. doi: 10.1111/papt.12197. Epub 2018 Sep 3. PMID 30175881
- [Background] Abu-Zidan FM, Abbas AK, Hefny AF. Clinical "case series": a concept analysis. Afr Health Sci. 2012 Dec;12(4):557-62. PMID 23515566
- [Background] Carey, T. A. (2008b). Perceptual control theory and the method of levels: Further contributions to a transdiagnostic perspective. International Journal of Cognitive Therapy, 1, 237-255.
- [Background] Carey TA, Mansell W, Tai SJ. A biopsychosocial model based on negative feedback and control. Front Hum Neurosci. 2014 Feb 28;8:94. doi: 10.3389/fnhum.2014.00094. eCollection 2014. PMID 24616685
- [Background] Carey, T.A. (2008). Hold That Thought! Two Steps to Effective Counselling and Psycho- therapy with the Method of Levels. Behavioural and Cognitive Psychotherapy, 37, 311-324
- [Background] Carey, T.A., Kelly, R.E., Mansell, W. & Tai, S. J. (2012). What's therapeutic about the therapeutic relationship? A hypothesis for practice informed by Perceptual Control Theory. The Cognitive Behaviour Therapist, 1-13.
- [Background] Churchman, A., Mansell, W., & Tai, S. (2019). A school-based feasibility study of method of levels: a novel form of client-led counselling. Pastoral Care in Education, 37(4), 331-346
- [Background] Cocklin AA, Mansell W, Emsley R, McEvoy P, Preston C, Comiskey J, Tai S. Client Perceptions of Helpfulness in Therapy: a Novel Video-Rating Methodology for Examining Process Variables at Brief Intervals During a Single Session. Behav Cogn Psychother. 2017 Nov;45(6):647-660. doi: 10.1017/S1352465817000273. Epub 2017 May 22. PMID 28528592
- [Background] First, M. B., Gibbon, M., Spitzer, R.L., & Williams, J. B. W. (2002). Structured Clinical interview for DSM-IV-TR axis 1 disorders (Research Version). New York: Biometrics Research Department, New York State Psychiatric Institute.
- [Background] Gaffney H, Mansell W, Tai S. Agents of change: Understanding the therapeutic processes associated with the helpfulness of therapy for mental health problems with relational agent MYLO. Digit Health. 2020 Mar 16;6:2055207620911580. doi: 10.1177/2055207620911580. eCollection 2020 Jan-Dec. PMID 32206331
- [Background] Griffiths R, Mansell W, Edge D, Carey TA, Peel H, J Tai S. 'It was me answering my own questions': Experiences of method of levels therapy amongst people with first-episode psychosis. Int J Ment Health Nurs. 2019 Jun;28(3):721-734. doi: 10.1111/inm.12576. Epub 2019 Jan 31. PMID 30701661